CLINICAL TRIAL: NCT07098936
Title: A Single-arm Phase II With safety-run-in Multicenter Study of Momelotinib in Patients With VEXAS Syndrome With or Without Associated Myelodysplastic Syndrome
Brief Title: Momelotinib in VEXAS Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-VEXAS-MMB
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: VEXAS Syndome; Myelo Dysplastic Syndrome
Keywords: VEXAS syndrome; Momelotinib; Myelodysplastic syndrome
MeSH Terms: conditions — VEXAS syndrome; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: a single-arm phase II with safety run-in study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Momelotinib treatment (Experimental): Patients will receive momelotinib.
  Interventions: Drug: Momelotinib treatment

INTERVENTIONS:
Drug: Momelotinib treatment — Patients included will receive momelotinib continuously until disease progression or loss of response, at physician's discretion.

SUMMARY:
Multicenter, phase II trial with safety run-in to evaluate the efficacy and safety of momelotinib in patients with VEXAS (Vacuoles, E1 enzyme, X-linked, Autoinflammatory and Somatic) syndrome with or without associated myelodysplastic syndrome (MDS).

The study will consist of two consecutive steps, a dose-finding safety run-in and a single-arm prospective phase II.

During safety run-in phase, three fixed dose levels will be tested according to a 3+3 design, using cohorts of size 3 in order to establish the maximum tolerated dose.

After this safety run-in phase, patients included in phase II will be treated with momelotinib at the maximum tolerated dose preliminary fixed.

Patients included in the phase II will receive momelotinib continuously until disease progression or loss of response, at physician's discretion.

All patients included in the study will receive glucocorticoids (prednisone/prednisolone equivalent) at baseline (at least > 10mg/day).

Response assessment regarding VEXAS related symptoms will be evaluated after 4, 12, 24 and 48 weeks. Response assessment regarding MDS features will be evaluated at 12 and 24 weeks.

DETAILED DESCRIPTION:
During safety run-in phase, the three fixed dose levels tested are :

* Dose level (DL) -1: 150 mg once daily (QD)
* DL1: 200 mg QD
* DL2: 300 mg QD. Between 6 and 18 patients will be enrolled during the safety run-in phase. Up to 39 patients could be included in the phase II study and will be treated with momelotinib at the maximum tolerated dose preliminary fixed during the safety run-in phase.

Baseline steroids daily dose required for VEXAS inflammatory manifestations will be defined during screening period (28 days period) for each patient. It is defined as the minimal daily dose of steroids used in the last 14 days prior momelotinib onset (according to physician disposition) that allow disease control. In case of related VEXAS inflammatory manifestation during screening period with a first fixed dose, an increased dose of steroids should be evaluated during at least an extra 14 days prior momelotinib onset. This baseline dose defined during screening period will be used for response criteria during follow-up.

Momelotinib treatment will be discontinued after 24 weeks at optimal dosing regimen (up to 300 mg/day), in case of absence of response.

Treatment might also be discontinued during follow-up in case of loss of response/hematological progression or non-tolerable adverse event.

ELIGIBILITY:
Inclusion Criteria:

* ECOG (Eastern Cooperative Oncology Group) performance status 0-2 at the time of screening
* Age ≥ 18 years
* Written informed consent
* Diagnosis of VEXAS (Vacuoles, E1 enzyme, X-linked, Autoinflammatory and Somatic) syndrome with UBA1 (Ubiquitin Like Modifier Activating Enzyme 1) mutation and clinically symptomatic disease requiring immunosuppressive treatment and at least 10mg/d of glucocorticoids
* Patients with uncontrolled symptoms related to VEXAS with prior treatment line(s) (including steroids)
* Patients refractory/dependent to steroids
* Single concomitant steroids therapy (e.g., prednisone or equivalent) at the time of inclusion is allowed
* For patients treated with other immunosuppressive/immunomodulatory therapy than glucocorticoids, a wash out period of 28 days is required prior momelotinib onset
* Erythropoietin/luspatercept used as a growth factor treatment is not allowed 28 days prior enrollment
* Adequate liver function (serum transaminases ≤ 3 x ULN (Upper Limits of Normal), Bilirubin ≤ 1.5 x ULN (isolated bilirubin > 1.5 x ULN is acceptable if bilirubin fractionated and direct bilirubin < 35%)
* Adequate renal function (creatinine clearance with MDRD (Modification of Diet in Renal Disease) formula > 30 ml/min)
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must:

  1. Have a negative serum or urine pregnancy test within 24 hours prior to beginning treatment on this study. Lactating patients are excluded.
  2. Agree to use, and to be able to comply with, effective contraception without interruption, 4 weeks before starting study drug throughout the entire duration study drug therapy (including doses interruptions) and for 12 weeks after the end of the study drug therapy.
  3. Agree to learn about the procedures for preservation of egg before starting treatment.
* Male patients must:

  1. Agree the need for the use of a condom if engaged in sexual activity with a woman of childbearing potential during the entire period of treatment, even if disruption of treatment and during 12 weeks after end of treatment.
  2. Agree to learn about the procedures for preservation of sperm before starting treatment.

Exclusion Criteria:

* Patients with MDS (Myelodysplastic syndrome) scheduled for allogeneic stem cell transplant or high risk MDS according to IWG (International Working Group) 2023
* Patients who are or have been already treated with Janus Kinase (JAK) inhibitors for VEXAS syndrome or another indication
* Patients who are unable to receive a starting daily dose of momelotinib of at least 100 mg
* Subjects with any other active malignancies are not eligible, except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which subject has been disease-free for at least 3 years
* Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 12 weeks prior to initiation of momelotinib
* Known infection with acute and chronic active Human Immunodeficiency Virus, Hepatitis B Virus, Hepatitis C Virus
* Any medical or psychiatric condition not allowing the informed consent of the subject
* Presence of clinically meaningful active bacterial, fungal, parasitic or viral infection which requires therapy
* Previous history of Progressive Multifocal Leuko-encephalopathy
* Active gastrointestinal conditions that may affect absorption
* No affiliation to a health insurance system
* Known hypersensitivity to the study investigational medicinal product, the metabolites, or formulation excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose of momelotinib | First 4-week cycle of momelotinib treatment
  The maximum tolerated dose (MTD) is defined by a target dose-limiting toxicities (DLT) rate of 30%, assessed during the observation window by a 3+3 design.
  The 3+3 design will enroll a first cohort of 3 patients at the starting dose of 200 mg/d:
  * If 0 of the 3 patients at the dose of 200 mg/d experienced a DLT during the first 4-week cycle of momelotinib, the dose will escalate to 300 mg/d for the next cohort.
  * If 1 of the 3 patients at the dose of 200 mg/d has a DLT, a cohort of three additional patients will be treated at the same dose of 200 mg/d.
  * If > 1 patient of the 3 patients at the dose of 200 mg/d have a DLT, the dose will de-escalate to 150 mg/d for the next cohort.
  The same process will be repeated until reaching the MTD. In total, between 6 and 18 patients will be enrolled during this safety run-in phase.
Clinical efficacy | During the 24 first weeks of momelotinib treatment
  Determination of overall clinical response rate at 24 weeks after momelotinib initiation on VEXAS related symptoms (including complete (CR) or partial response (PR)) :
  * CR includes complete disappearance of symptoms related to systemic inflammation according to treating physician and daily dose of steroids ≤ 10 mg/d (equivalent prednisolone).
  * PR includes complete disappearance of symptoms related to systemic inflammation according to treating physician and reduction of at least 50% of daily dose steroids compared to baseline and/or daily dose of steroids > 10 mg/d.

SECONDARY OUTCOMES:
Pharmacokinetic | At cycle 1 Day 8-9 and cycle 13 Day 8-9
  Concentrations of momelotinib and its major metabolite M21 will be determined in plasma samples using the currently approved bioanalytical methodology by Frontage Laboratories Inc.
  Pharmacokinetic sampling will be only performed for patients in safety run-in phase.
  Samples should be obtained at cycle 1 Day 8 and cycle 13 Day 8, at times following : Pre-dose then at 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8h and at 24 h post Day 8 dose.
Incidence of Treatment-Emergent Adverse Events | From enrollment to the end of treatment at 48 weeks
  Collection of Adverse events (AE), serious AE (SAE) and toxicities as measured by NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) v5.0
Response | After 4, 12, 24 and 48 weeks of momelotinib treatment
  Determination of overall clinical response rates (including Complete Response or Partial Response) and biological response rates (complete or partial)
Hematological response | After 16 weeks of momelotinib treatment
  Erythroid hematological improvement will be assessed by the investigators according to IWG 2018 criteria through collection of transfusion records and hematology parameters.
Steroids dose reduction | After 24 weeks of momelotinib treatment
  Steroids dose reduction compared to baseline and/or steroids withdrawal rates
Overall survival | From enrollment to the end of treatment at 12 months
  Overall survival assessment
Myelodysplastic syndrome (MDS) evolution | From baseline at 12 and 24 weeks of momelotinib treatment
  Changes in the underlying MDS from baseline, at 12 and 24 weeks, including MDS progression based on hematological, cytogenetic and molecular analysis
Duration of response | From enrollment to the end of treatment at 48 weeks
  Duration of response on VEXAS symptoms defined as the time from the date of initial documentation of a clinical response (Complete Response or Partial Response) to the date of first documented evidence of relapse or death
Best clinical response | From enrollment to the end of treatment at 48 weeks
  Determination of time to the first and best clinical response
RBC independency | From enrollment to the end of treatment at 48 weeks
  Duration of Red Blood Count (RBC) independency in patients with RBC dependency at time of inclusion, according to IWG 2018 criteria
UBA1 VAF | From enrollment to the end of treatment at 24 weeks
  Evolution of UBA1 (Ubiquitin Like Modifier Activating Enzyme 1) VAF (Variant Allelic Frequency) from baseline to W4, W12 and W24 after momelotinib treatment

OTHER OUTCOMES:
Validation of the VEXAS personal scoring system (VPSS) | After 4, 12 and 24 weeks of momelotinib treatment
  Measurement of VPSS to validate the score currently under development which would allow objectively quantifying the impact of VEXAS-related symptoms on patients' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Maël HEIBLIG, MD, Principal Investigator — CH Lyon Sud
Locations (11):
- France (11):
  - CHU d'Angers - Service des Maladies du sang, Angers
  - CHU Estaing - Service d'Hématologie Clinique, Clermont-Ferrand
  - Hôpital Claude Huriez - Service de Médecine Interne, Lille
  - CHU Nantes - Hôtel Dieu - Service d'Hématologie Clinique, Nantes
  - Hôpital Saint Louis - Service hématologie séniors, Paris
  - Hôpital Saint-Antoine - Service de Médecine Interne, Paris
  - CHU de Haut-Lévèque - Centre F. Magendie - Service des Maladies du sang, Pessac
  - CH Lyon sud - Service d'Hématologie Clinique, Pierre-Bénite
  - Hôpital Pontchaillou Service d'hématologie clinique et service de médecine interne, Rennes
  - IUCT Oncopole Département d'hématologie / Unité de médecine interne, Toulouse
  - CHU de Tours - Hôpital Bretonneau - Service de Médecine Interne, Tours

IPD SHARING:
Plan to Share IPD: No